CLINICAL TRIAL: NCT03027687
Title: Effects of Repetitive tDCS on ad Libitum Smoking Behavior: An EMA and EEG Study
Brief Title: Effects of Repetitive tDCS on ad Libitum Smoking Behavior: EMA and EEG Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Ingmar Franken, Prof. Dr., Erasmus Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NL58190.078.16
Record Dates: First submitted 2017-01-05; First posted 2017-01-23 (Estimated); Last update posted 2018-11-16 (Actual); Status verified 2018-11

CONDITIONS: Addiction
Keywords: Smoking; EMA; ERPs; tDCS; Cigarette consumption; Inhibitory control; Reward processing; Tobacco addiction; Craving; electrophysiological
MeSH Terms: conditions — Behavior, Addictive; Smoking | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Real transcranial Direct Current Stimulation (Experimental): This group will receive bilateral tDCS (left cathodal/right anodal) over the DLPFC. The stimulation will take place two times daily for 13 minutes with a rest interval of 20 minutes for three days in one week.
  Interventions: Device: tDCS
- Sham tDCS (Sham Comparator): The control group receives sham, for which the stimulator will be gradually turned off after 30 seconds.
  Interventions: Device: tDCS

INTERVENTIONS:
Device: tDCS — tDCS is an electrical brain stimulation method
  Other Names: transcranial direct current stimulation

SUMMARY:
Bilateral (left cathodal/ right anodal) transcranial Direct Current Stimulation (tDCS) over the dorsolateral prefrontal cortex (DLPFC) seems to reduce craving and to increase the time till smoking the first cigarette after the intervention. The current study explores whether actual cigarette consumption decreases after repetitive tDCS. Cigarette consumption and craving will therefore be measured by means of EMA, before (at baseline), during and after multiple tDCS sessions, and at 3 months follow-up.

To study the working mechanism behind the effects of tDCS, electrophysiological responses (ERPs) and behavioral measures of cognitive control functioning will be taken into account at baseline, one day after the last tDCS session and at three months follow up.

We hypothesize that cigarette consumption will decrease after repetitive tDCS, and that this effect is associated with better cognitive control functioning.

DETAILED DESCRIPTION:
The proposed experiment is a double-blind randomized placebo-controlled trial. 60 smokers will be randomly assigned to two conditions, namely tDCS or sham (placebo).

Participants will receive real tDCS or sham for three days in one week. The interventions contain twice daily sessions for 13 minutes with an interval of 20 min. Moreover, on the first treatment day and the day after the treatment week, participants complete a number of questionnaires, and perform two psychological tasks (a gambling task and the Go/NoGo task) to measure cognitive control functioning (e.g. risky decision making and inhibitory control respectively). During these tasks, event-related potentials will be recorded by means of EEG. After three months, participants are asked to return to fill out the same questionnaires and perform the same psychological tasks as before, to measure the lasting effect of tDCS. During this last session, event-related potentials will also be recorded. In addition, carbon monoxide levels will be measured on all days where subjects perform the tasks.

EMA:

For three weeks, starting the week before tDCS treatment, participants are asked to log every cigarette before they smoke one. During these weeks, participants complete EMA questionnaires on their mobile phone about cigarette consumption, craving, and affect that will take approximately 5 minutes. The EMA questionnaire will be presented four times daily on a quasi-random basis. Finally, during end-of-day assessments participants have the possibility to indicate any missed cigarettes. At three months follow-up, participants are asked to undergo the same EMA procedure for one more week, to study the lasting effects of tDCS.

ELIGIBILITY:
Inclusion Criteria:

* Currently smoking 10 or more cigarettes a day
* The ability to speak, read, and write in Dutch at an eight-grade literacy level

Exclusion Criteria:

* The current abuse of a substance other than nicotine or caffeine
* History of neurological or psychiatric disorders
* Any contraindication for electrical brain stimulation procedures such as electronic implants or metal implants
* Pregnancy or breast-feeding
* In the process of quitting smoking

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Mean number of cigarettes a day at 3 months follow up | 3 months
  The mean number of cigarettes will be measured at three months follow-up by means of Ecological Momentary Assessments (EMA). This means that participants are asked to report every cigarette they smoke at the moment they're about to smoke it with an app on their mobile phone. Participants do this during the week before the last EEG session at three months follow-up.The mean number will be calculated over this week

SECONDARY OUTCOMES:
Mean number of cigarettes a day one week after tDCS | 1 week
  The mean number of cigarettes will be measured at one week after the last tDCS session by means of Ecological Momentary Assessments (EMA). This means that participants are asked to report every cigarette they smoke at the moment they're about to smoke it with an app on their mobile phone. Participants do this for one week starting from the last tDCS session. The mean number will be calculated over this week
Craving at 3 months follow-up | 3 months
  Participants receive 4 prompts a day in the app on the smartphone to fill out questions about craving for 1 week starting the week before the last EEG session at three months follow-up
Affect 3 months after tDCS | 3 months
  Participants receive 4 prompts a day in the app on the smartphone to fill out questions about affect for 1 week starting the week before the last EEG session at three months follow-up
Craving one week after tDCS | 1 week
  Participants receive 4 prompts a day in the app on the smartphone to fill out questions about craving for 1 week starting the day after the last tDCS session
Affect one week after tDCS | 1 week
  Participants receive 4 prompts a day in the app on the smartphone to fill out questions about affect for 1 week starting the day after the last tDCS session
Behavioral responses of risk-taking | 3 times: at baseline, one day after all tDCS sessions, and at 3 months follow-up
  Measured with the two-choice gambling task: proportion of high-risk (higher values) choices
Behavioral responses of inhibitory control | 3 times: at baseline, one day after all tDCS sessions, and at 3 months follow-up
  Measured by proportion correctly inhibited NoGo trials on the Go/NoGo task
Feedback Related Negativity (FRN): Event Related potential (ERP) of reward processing | 3 times: at baseline, one day after all tDCS sessions, and at 3 months follow-up
  Measured with the two choice gambling task. After the choice (high/low risk) is made, participants receive feedback (either they lose or win). The Feedback Related Negativity (FRN) will be measured after feedback by means of EEG.
Reward related P300: Event related potential (ERP) of reward processing | 3 times: at baseline, one day after all tDCS sessions, and at 3 months follow-up
  Measured with the two choice gambling task. After the choice (high/low risk) is made, participants receive feedback (either they lose or win). The reward related P300 will be measured 300-500 ms after feedback by means of EEG.
N200: Event related potential (ERP) of inhibitory control | 3 times: at baseline, one day after all tDCS sessions, and at 3 months follow-up
  The N200 will be measured after NoGo trials in the Go/NoGo task
P300: Event related potential (ERP) of inhibitory control | 3 times: at baseline, one day after all tDCS sessions, and at 3 months follow-up
  The P300 will be measured after NoGo trials in the Go/NoGo task
Error related negativity: Event related potential (ERP) of error processing | 3 times: at baseline, one day after all tDCS sessions, and at 3 months follow-up
  Wrong responses to Go and NoGo trials in the Go/NoGo task will be used to assess the error related negativity (ERN)
Course of cigarette consumption | 2 weeks
  Number of cigarettes (and craving) a day starting on the first tDCS day until one week after the last tDCS intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Erasmus University, Rotterdam, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Verveer I, Remmerswaal D, van der Veen FM, Franken IHA. Long-term tDCS effects on neurophysiological measures of cognitive control in tobacco smokers. Biol Psychol. 2020 Oct;156:107962. doi: 10.1016/j.biopsycho.2020.107962. Epub 2020 Sep 23. PMID 32979429
- [Derived] Verveer I, Remmerswaal D, Jongerling J, van der Veen FM, Franken IHA. No effect of repetitive tDCS on daily smoking behaviour in light smokers: A placebo controlled EMA study. PLoS One. 2020 May 22;15(5):e0233414. doi: 10.1371/journal.pone.0233414. eCollection 2020. PMID 32442205